CLINICAL TRIAL: NCT04091516
Title: The Feasibility, Implementation and Efficacy of a Plant-Based Weight-Loss Program in a Practice-Based Setting
Brief Title: Feasibility & Implementation of a Plant-Based Weight-Loss Program in an Office-Based Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00037092
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Weight Loss; Blood Pressure; Lipid Disorder; PreDiabetes; Diabete Mellitus
Keywords: weight loss; body composition; lipids; hemoglobin A1c; blood pressure
MeSH Terms: conditions — Weight Loss; Lipid Metabolism Disorders; Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Prospective interventional study without a control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-fat plant-based diet (Other): For 12 weeks, participants will follow a diet comprised of whole grains, vegetables, legumes, and fruits, with no restriction on energy intake. Animal products and added oils will be excluded. Except for light refreshments and tastings at the group sessions, no meals will be provided. Participants will handle their own food preparation and purchases, with guidance from the education team, with no restriction on energy intake.
  Interventions: Behavioral: Low-fat plant-based diet

INTERVENTIONS:
Behavioral: Low-fat plant-based diet — Participants will follow a diet that consists of whole grains, vegetables, legumes, and fruits, with no restriction on energy intake. Animal products and added oils will be excluded. Except for light refreshments and tastings at the group sessions, no meals will be provided. Participants will handle their own food preparation and purchases, with guidance from the education team, with no restriction on energy intake.

SUMMARY:
This prospective study aims to assess the feasibility and implementation of a plant-based, weight-loss program in an office setting. The study will also assess changes in body weight, blood pressure, plasma lipids, glycated hemoglobin, and body composition with a 12-week, plant-based, weight-loss program. These health benefits may illustrate feasibility to physicians and healthcare professionals elsewhere.

DETAILED DESCRIPTION:
This will be a prospective interventional study to evaluate the feasibility, implementation and efficacy of 12-week plant-based, weight-loss program that is carried out in an office setting and is open to participation to the general public via local print and online advertising or whichever methods apply. The program will include weekly education and support, and assessment of blood pressure, lipids, hemoglobin A1c, and body composition before and after starting the program. The price of the program, $645, will cover the costs of weekly education, blood pressure check, laboratory testing and body composition analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥18 years of age

Exclusion Criteria:

* Use of recreational drugs in the past 6 months
* Pregnancy or intention to become pregnant during the study period, as verified by self-report
* Unstable medical or psychiatric illness
* Lack of English fluency
* Inability to maintain current medication regimen
* Inability or unwillingness to participate in all components of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | Change from baseline to 12 weeks
  With participants wearing light, indoor clothing but without shoes, body weight will be measured to the nearest 0.1 kg, using a digital scale. Body weight will also be assessed at each weekly session, but only data from the week 1 (pre-program) and week 12 (post-program) will be included in the analysis.

SECONDARY OUTCOMES:
Blood pressure | Change from baseline to 12 weeks
  Blood pressure will be measured using an automated oscillometric device.
Plasma cholesterol and triacylglycerol concentrations | Change from baseline to 12 weeks
  Will be measured using standard methods.
hemoglobin A1c | Change from baseline to 12 weeks
  will be measured using standard methods.
Body Composition | Change from baseline to 12 weeks
  Body composition will be measured by dual energy x-ray absorptometry (Lunar iDXA, GE Healthcare; Madison, WI) with Encore® 2005 v.9.15.010 software. The iDXA can measure body composition with low x-ray exposure and short scanning time. The iDXA unit will be calibrated daily using the GE Lunar calibration phantom, and a trained operator will perform all scans following standard protocol for participant positioning. The iDXA is equipped with the CoreScan module (GE Healthcare, Madison, WI), which can also provide an estimate of visceral adipose tissue volume and mass.

CONTACTS AND LOCATIONS:
Overall Officials: Vanita J Rahman, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Barnard Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will make individual data available to other researchers upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 31, 2020
Access Criteria: Will make study data available upon request

REFERENCES:
- [Background] Tonstad S, Butler T, Yan R, Fraser GE. Type of vegetarian diet, body weight, and prevalence of type 2 diabetes. Diabetes Care. 2009 May;32(5):791-6. doi: 10.2337/dc08-1886. Epub 2009 Apr 7. PMID 19351712
- [Background] Barnard ND, Levin SM, Yokoyama Y. A systematic review and meta-analysis of changes in body weight in clinical trials of vegetarian diets. J Acad Nutr Diet. 2015 Jun;115(6):954-69. doi: 10.1016/j.jand.2014.11.016. Epub 2015 Jan 22. PMID 25620754
- [Background] Barnard N, Scherwitz L, Ornish D. Adherence and acceptability of a lowfat vegetarian diet among patients with cardiac disease. J Cardiopulmonary Rehabil 1992;12:423-31
- [Background] Barnard N, Scialli A, Bertron P, Hurlock D, Edmonds K. Acceptability of a therapeutic low-fat, vegan diet in premenopausal women. J Nutr Educ 2000;32:314-9.
- [Background] American Dietetic Association; Dietitians of Canada. Position of the American Dietetic Association and Dietitians of Canada: Vegetarian diets. J Am Diet Assoc. 2003 Jun;103(6):748-65. doi: 10.1053/jada.2003.50142. PMID 12778049
- [Background] Barnard ND, Scialli AR, Turner-McGrievy G, Lanou AJ. Acceptability of a low-fat vegan diet compares favorably to a step II diet in a randomized, controlled trial. J Cardiopulm Rehabil. 2004 Jul-Aug;24(4):229-35. doi: 10.1097/00008483-200407000-00004. PMID 15286527
- [Background] Barnard ND, Gloede L, Cohen J, Jenkins DJ, Turner-McGrievy G, Green AA, Ferdowsian H. A low-fat vegan diet elicits greater macronutrient changes, but is comparable in adherence and acceptability, compared with a more conventional diabetes diet among individuals with type 2 diabetes. J Am Diet Assoc. 2009 Feb;109(2):263-72. doi: 10.1016/j.jada.2008.10.049. PMID 19167953
- [Background] Barnard ND, Akhtar A, Nicholson A. Factors that facilitate compliance to lower fat intake. Arch Fam Med. 1995 Feb;4(2):153-8. doi: 10.1001/archfami.4.2.153. PMID 7842153
- [Background] Becker M. The health belief model and personal health behavior. Health Education Monographs 1974;2:324-473.
- [Background] U.S. Census Bureau. Quick Facts. District of Columbia. Internet: http://www.census.gov/quickfacts/table/RHI125215/11, accessed August 22, 2016.